CLINICAL TRIAL: NCT00269685
Title: Comparative Prospective Study of Vasopressin and Catecholamine in Septic Shock
Brief Title: Comparison of Vasopressin and Other Pressors in Septic Shock
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-33-R2
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2006-05-29 (Estimated); Status verified 2005-08

CONDITIONS: Shock, Septic
Keywords: Septic shock; catecholamine; vasopressin; tonometria; lactate
MeSH Terms: conditions — Shock, Septic; Diabetes Insipidus | interventions — Vasopressins

INTERVENTIONS:
Drug: vasopressin

SUMMARY:
The purpose of this study is to compare the classical tactics in the treatment of septic shock (dopamine, noradrenalin and dobutamine) to the use of vasopressin as first choice pressor.

Vasopressin seems to be an interesting alternative in the treatment of septic shock. To this date, available studies have showed that it could correct hyperkinetic syndrome and vasoplegia in septic shocks without noticeable side effect. It as been demonstrated that vasopressin improves renal function, as no effect on digestive organs and as no metabolic effect.

ELIGIBILITY:
Inclusion Criteria:

* Legally major patient presenting a septic shock.

The time window between beginning of symptoms and onset of treatment is established at 12 hours.

The patient must be intubated and mechanically ventilated.

Patient presenting a mean arterial blood pressure of less than 60 mm Hg after adequate fluid resuscitation (at least 1 L of colloid or crystalloid) and 10 ug/Kg/min of dopamine.

Patient presenting a cardiac index of at least 3 L/min/m2

Exclusion Criteria:

* Shock other than septic
* cardiac hypokinesia
* a pre-existing organic renal failure that needs hemodyalisis
* oesophagal or gastric phatology that would lead to a naso-gastric tube contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2000-07

PRIMARY OUTCOMES:
To compare the efficiency of vasopressine to the standard and usual treatment of septic shock on the reverse of the hemodynamic criterion of septic shock

SECONDARY OUTCOMES:
To compare these two categories of treatment on:
tonometric parameters
renal function
in term of tolerance: metabolic effects (increase in lactate and glycaemia), cardiac effects (tachycardia being defined as a heart rate increase of 15%), increase of cardiac enzymes (troponine, CK, CK-MB), and cutanuous vasoconstriction.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lesur, Ph d, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke

REFERENCES:
- [Background] American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference: definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. Crit Care Med. 1992 Jun;20(6):864-74. PMID 1597042
- [Background] Landry DW, Levin HR, Gallant EM, Ashton RC Jr, Seo S, D'Alessandro D, Oz MC, Oliver JA. Vasopressin deficiency contributes to the vasodilation of septic shock. Circulation. 1997 Mar 4;95(5):1122-5. doi: 10.1161/01.cir.95.5.1122. PMID 9054839
- [Background] Luk J, Ajaelo I, Wong V, Wong J, Chang D, Chou L, Reid IA. Role of V1 receptors in the action of vasopressin on the baroreflex control of heart rate. Am J Physiol. 1993 Sep;265(3 Pt 2):R524-9. doi: 10.1152/ajpregu.1993.265.3.R524. PMID 8214142
- [Background] Malay MB, Ashton RC Jr, Landry DW, Townsend RN. Low-dose vasopressin in the treatment of vasodilatory septic shock. J Trauma. 1999 Oct;47(4):699-703; discussion 703-5. doi: 10.1097/00005373-199910000-00014. PMID 10528604
- [Background] Reid IA. Role of vasopressin deficiency in the vasodilation of septic shock. Circulation. 1997 Mar 4;95(5):1108-10. doi: 10.1161/01.cir.95.5.1108. No abstract available. PMID 9054835
- [Background] Rozenfeld V, Cheng JW. The role of vasopressin in the treatment of vasodilation in shock states. Ann Pharmacother. 2000 Feb;34(2):250-4. doi: 10.1345/aph.19066. PMID 10676834